CLINICAL TRIAL: NCT00190385
Title: Screening of Hepatocellular Carcinoma in Patients With Compensated Cirrhosis. A Randomized Trial Comparing Two Periodicities of Ultrasonographic Surveillance: 3-month vs 6-month
Brief Title: Screening of Hepatocellular Carcinoma in Patients With Compensated Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); UNICANCER (Other)
Responsible Party: Sylla KHAOUSSOU, Department of Clinical Research of developpement
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: AOM03009
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2007-03

CONDITIONS: Compensated Cirrhosis
Keywords: Cirrhosis; Hepatocellular carcinoma; Screening; Randomized; HBV; HCV; alcohol; hemochromatosis
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular; Hemochromatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator)
  Interventions: Procedure: Ultrasonographic screening

INTERVENTIONS:
Procedure: Ultrasonographic screening — Ultrasonographic screening

SUMMARY:
Liver carcinoma is becoming the main complication of cirrhosis. Treatment of symptomatic or large tumors is disappointing. Regular ultrasonographic screening of small (curable) tumors is currently recommended, but the best periodicity is unknown.This randomized trial is aimed to compare 6-month (current recommendation) and 3-month ultrasonographic screenings.

DETAILED DESCRIPTION:
Patients: All consecutive patients with compensated HBV, HCV, alcohol or hemochromatosis-related cirrhosis (without any previous clinical complication including liver cancer).

Randomization: factorial: ultrasonography (3-month versus 6-month); serum alfa-fetoprotein assay (none versus 6-month).

End points: rate of small tumors (first main criteria); survival (second main criteria).

ELIGIBILITY:
Inclusion Criteria:

* Compensated cirrhosis

Exclusion Criteria:

* Antecedent of osmic acid synoviorthesis or of isotopic synoviorthesis of the studied knee
* Intra-articular injection of triamcinolone hexacetonide in three months preceding the inclusion or by a different corticoid in the month preceding the inclusion
* Evolutionary infectious or neoplastic pathology

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2000-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence of small hepatocellular carcinoma (HCC) | 6 months versus 3 months

SECONDARY OUTCOMES:
Survival | during the study
Clinical value of serum alfa-fetoprotein assay | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Trinchet, Pr, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Jean Verdier, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Ganne-Carrie N, Nahon P, Chaffaut C, N'Kontchou G, Layese R, Audureau E, Chevret S; CIRRAL group; ANRS CO12 CirVir group. Impact of cirrhosis aetiology on incidence and prognosis of hepatocellular carcinoma diagnosed during surveillance. JHEP Rep. 2021 Mar 26;3(3):100285. doi: 10.1016/j.jhepr.2021.100285. eCollection 2021 Jun. PMID 34522876
- [Derived] Nery F, Chevret S, Condat B, de Raucourt E, Boudaoud L, Rautou PE, Plessier A, Roulot D, Chaffaut C, Bourcier V, Trinchet JC, Valla DC; Groupe d'Etude et de Traitement du Carcinome Hepatocellulaire. Causes and consequences of portal vein thrombosis in 1,243 patients with cirrhosis: results of a longitudinal study. Hepatology. 2015 Feb;61(2):660-7. doi: 10.1002/hep.27546. Epub 2015 Jan 5. PMID 25284616
- [Derived] Trinchet JC, Chaffaut C, Bourcier V, Degos F, Henrion J, Fontaine H, Roulot D, Mallat A, Hillaire S, Cales P, Ollivier I, Vinel JP, Mathurin P, Bronowicki JP, Vilgrain V, N'Kontchou G, Beaugrand M, Chevret S; Groupe d'Etude et de Traitement du Carcinome Hepatocellulaire (GRETCH). Ultrasonographic surveillance of hepatocellular carcinoma in cirrhosis: a randomized trial comparing 3- and 6-month periodicities. Hepatology. 2011 Dec;54(6):1987-97. doi: 10.1002/hep.24545. PMID 22144108